CLINICAL TRIAL: NCT00799864
Title: A Phase II, Open Label, Single Arm Trial to Evaluate the Pharmacokinetics,Safety, Tolerability, and Antiviral Activity of Rilpivirine (TMC278) in Antiretroviral Naive HIV-1 Infected Adolescents and Children Aged >= 6 to <18 Years
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, Tolerability, and Antiviral Activity of Rilpivirine (TMC278) in Human Immunodeficiency Virus Infected Adolescents and Children Aged Greater Than or Equal to 6 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002677; TMC278-TiDP38-C213 (Other: Janssen Sciences Ireland UC); 2008-001696-30 (EudraCT Number)
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: HIV-1
Keywords: HIV Infection; Antiretroviral; HIV-1; AIDS; Children; Rilpivirine (TMC278); Pediatric
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Rilpivirine; Zidovudine; abacavir; Tenofovir; Lamivudine; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Rilpivirine (TMC278) (Experimental): The patients received rilpivirine with 2 nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) as a background regimen in cohort 1 [aged greater than or equal to (> =) 12 to less than (<) 18 years] for up to 240 weeks which is already completed and recruitment closed and will receive this treatment in cohort 2 (children aged > = 6 to < 12 years) for up to 48 weeks. The NRTIs include zidovudine, abacavir, or tenofovir disoproxil fumarate in combination with lamivudine or emtricitabine.
  Interventions: Drug: Rilpivirine; Drug: Zidovudine; Drug: Abacavir; Drug: Tenofovir disoproxil fumarate; Drug: Lamivudine; Drug: Emtricitabine

INTERVENTIONS:
Drug: Rilpivirine — Patients will receive rilpivirine (RPV) tablet 25 milligram dose or an adjusted dose orally once daily in Cohort 1 (adolescents aged >=12 to <18 years) up to 240 weeks. Patients will receive RPV weight-adjusted dose orally once daily in Cohort 2 (children aged >=6 to <12 years) or 25 mg once daily for up to 48 weeks.
Drug: Zidovudine — Type=exact, form= appropriate pediatric formulation, unit=mg, route=oral. The patients may receive this selected NRTI together with another NRTI once daily for up to 48 weeks (Cohort 2) and 240 weeks (Cohort 1).
Drug: Abacavir — Type=exact, form=appropriate pediatric formulation, unit=mg, route=oral. The patients may receive this selected NRTI together with another NRTI once daily for up to 48 weeks (Cohort 2) and 240 weeks (Cohort 1).
Drug: Tenofovir disoproxil fumarate — Type=exact, form=appropriate pediatric formulation, unit=mg, route=oral. The patients may receive this selected NRTI together with another NRTI once daily for 240 weeks (Cohort 1).
Drug: Lamivudine — Type=exact, form=appropriate pediatric formulation, unit=mg, route=oral. The patients may receive this selected NRTI together with another NRTI once daily for up to 48 weeks (Cohort 2) and 240 weeks (Cohort 1).
Drug: Emtricitabine — Type=exact, form=appropriate pediatric formulation, unit=mg, route=oral. The patients may receive this selected NRTI together with another NRTI once daily for up to 48 weeks (Cohort 2) and 240 weeks (Cohort 1).

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety and antiviral activity of rilpivirine (TMC278) 25 milligram (mg) or adjusted dose once daily in combination with an investigator-selected background regimen containing 2 nucleoside/nucleotide reverse transcriptase inhibitors (N[t]RTIs) (zidovudine [AZT], abacavir [ABC], or tenofovir disoproxil fumarate [TDF] in combination with lamivudine [3TC] or emtricitabine [FTC] in antiretroviral (ARV) treatment-naïve adolescents and children aged greater than or equal to (>=) 6 to less than (<) 18 years.

DETAILED DESCRIPTION:
This is a Phase II, open-label (all people involved know the identity of the assigned drug) and single arm study. The study will consist of a screening period of maximum 8 weeks, an initial treatment period of 48 weeks, a post week 48 treatment extension period of 4 years (Cohort 1 only), and a 4 week follow-up (cohort 2 only) period. Participants who withdraw from the trial on or before the Week 48 visit or subjects with ongoing (serious) adverse events ([S]AEs), laboratory abnormalities, or viral load increase at the last on-treatment visit in the extension, will be seen for a follow-up visit 4 weeks later. The initial 48-week treatment period will be structured into 2 age Cohorts; Cohort 1 (Aged greater than or equal to [>=] 12 to less than [<] 18 years) and Cohort 2 (Children Aged >= 6 to < 12 years). The trial is designed to evaluate the steady-state pharmacokinetic (PK) profile (based on intensive PK analysis) and the short-term safety and antiviral activity of rilpivirine (RPV). Participants will receive RPV 25 milligram (mg), or weight-adjusted dose orally once daily for 240 weeks when administered in combination with 2 nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs). The trial will also evaluate long-term (48 weeks and 240 weeks [Cohort 1]) safety, efficacy, and pharmacokinetics of rilpivirine in combination with the background regimen of 2 NRTIs. Patients safety will be monitored throughout the study and during the follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Has documented human immuno deficiency virus (HIV-1) infection
* Patients who meet the following criteria; a) Cohort 1: Patients Aged greater than or equal to (>=) 12 to less than (<) 18 years, weight is >= 32 kilogram (kg), b) Cohort 2; Aged >= 6 to < 12 years, weight is >= 17 kg
* Must have HIV-1 plasma viral load at screening greater than equal to 500 HIV-1 ribonucleic acid (RNA) copies/mL
* Have not received treatment with a therapeutic HIV vaccine or an HIV drug with the exception of a single dose of nevirapine (NVP) (Cohort 1 and Cohort 2) or up to 6 weeks of zidovudine (AZT) use (Cohort 2 only) prior to screening to prevent mother-to-child transmission (MTCT)
* In the judgment of the investigator, it is appropriate to initiate antiretroviral therapy (ARV) therapy based on a patient's medical condition and taking into account guidelines for the treatment of HIV-1 infection in children of this age group

Exclusion Criteria:

* Any previous use of ARVs with the exception of single dose NVP (Cohort 1 and Cohort 2) or up to 6 weeks of AZT (Cohort 2 only) to prevent MTCT
* Plasma viral load at screening greater than 100,000 HIV-1 RNA copies/mL
* Documented genotypic evidence of non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance at screening or from historical data available in the source documents
* Use of disallowed concomitant therapy from 4 weeks prior to the baseline visit
* Patient has any currently active Acquired Immunodeficiency Syndrome (AIDS) defining illness
* Patient has active tuberculosis and/or is being treated for tuberculosis at screening
* Personal history of cardiac disease (including congenital heart disease), or symptomatic arrhythmias, with the exception of sinus arrhythmia; personal history of asymptomatic arrhythmias is excluded if the asymptomatic arrhythmia is clinically significant in the opinion of the investigator

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (17):
- United States (2):
  - Syracuse, New York
  - Memphis, Tennessee
- India (2):
  - Chennai
  - Mangalore
- Nairobi, Kenya
- Bucharest, Romania
- South Africa (6):
  - Bloemfontein
  - Dundee
  - Middelburg
  - Pretoria
  - Thabazimbi
  - Vosloorus
- Thailand (2):
  - Bangkok
  - Nonthaburi
- Uganda (2):
  - Entebbe
  - Kampala
- Kiev, Ukraine

REFERENCES:
- [Derived] Lombaard J, Ssali F, Thanyawee P, Fourie J, Vanveggel S, Linthicum C, Van Eygen V, Van Solingen-Ristea R. Phase 2 Open-Label Study of Long-Term Safety, Tolerability, and Antiviral Activity of Rilpivirine in Antiretroviral-Naive Adolescents Living with HIV-1. Antimicrob Agents Chemother. 2022 Feb 15;66(2):e0091621. doi: 10.1128/AAC.00916-21. Epub 2021 Dec 6. PMID 34871089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 54 antiretroviral-naïve human Immunodeficiency Virus-1 (HIV-1) infected adolescents (aged greater than or equal to [>=] 12 to less than [<] 18 years) and children (aged >=6 to <12 years) were enrolled and treated in Cohort 1 and Cohort 2, respectively.
Pre-assignment Details: As of Protocol Amendment 10 (PA 10), for Cohort 2 children >=6 to <12 years of age, post Week 48 treatment extension period of 4 years was removed. Hence, the planned efficacy analysis were performed till Week 48 only whereas safety analysis was performed and reported up to Week 240.
Groups:
- Cohort 1 Adolescents: Rilpivirine 25 mg: Adolescents (aged >=12 to <18 Years) received rilpivirine (RPV) tablet 25 mg orally QD up to 240 weeks in combination with an investigator-selected background regimen containing 2 nucleos(t)ide reverse transcriptase inhibitors (N[t]RTIs) (zidovudine [AZT], abacavir [ABC] or tenofovir disoproxil fumarate [TDF] in combination with lamivudine [3TC] or emtricitabine [FTC].
- Cohort 2 Children (>=25 kg): Rilpivirine 25 mg: Children (aged >=6 to <12 years) with body weight >=25 kg received rilpivirine 25 mg tablet orally QD from Day 1 up to 240 weeks (for participants recruited up to protocol amendment 9); up to 48 weeks (for participants recruited after implementation of protocol amendment 10) in combination with an investigator-selected background regimen containing 2 N[t]RTIs: AZT, ABC, or TDF in combination with 3TC or FTC.
- Cohort 2 Children (<25 kg): Rilpivirine 25 mg: Children (aged >=6 to <12 years) with body weight <25 kg received rilpivirine 25 mg tablet orally QD from Day 1 up to 240 weeks (for participants recruited up to protocol amendment 9); up to 48 weeks (for participants recruited after implementation of protocol amendment 10) in combination with an investigator-selected background regimen containing 2 N[t]RTIs: AZT, ABC, or TDF in combination with 3TC or FTC.
- Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg: Children (aged >=6 to <12 years) with body weight >=20 to <25 kg received rilpivirine 15 mg (6 tablets of 2.5 mg) orally QD from Day 1 up to 240 weeks (for participants recruited up to protocol amendment 9); up to 48 weeks (for participants recruited after implementation of protocol amendment 10) in combination with an investigator-selected background regimen containing 2 N[t]RTIs: AZT, ABC, or TDF in combination with 3TC or FTC.
- Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg: Children (aged >=6 to <12 years) with body weight <20 kilograms (kg) received rilpivirine 12.5 mg (5 tablets of 2.5 mg) orally QD from Day 1 up to 240 weeks (for participants recruited up to protocol amendment 9); up to 48 weeks (for participants recruited after implementation of protocol amendment 10) in combination with an investigator-selected background regimen containing 2 N[t]RTIs: AZT, ABC, or TDF in combination with 3TC or FTC.
Period: Overall Study
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 Children (>=25 kg): Rilpivirine 25 mg | Cohort 2 Children (<25 kg): Rilpivirine 25 mg | Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg | Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg
Started | 36 | 9 | 5 | 2 | 2
Completed | 25 | 6 | 3 | 2 | 2
Not Completed | 11 | 3 | 2 | 0 | 0
Not completed — Participant reached a virologic endpoint | 9 | 2 | 2 | 0 | 0
Not completed — Other | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 Children (>=25 kg): Rilpivirine 25 mg | Cohort 2 Children (<25 kg): Rilpivirine 25 mg | Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg | Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg | Total
Number analyzed (Participants) | 36 | 9 | 5 | 2 | 2 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.66) | 9.4 (1.67) | 9.2 (0.84) | 6.5 (0.71) | 6 (0) | 12.6 (3.29)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 9 | 5 | 2 | 2 | 18
  Adolescents (12-17 years) | 36 | 0 | 0 | 0 | 0 | 36
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 0 | 0
  From 65 to 84 years | 0 | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 3 | 2 | 1 | 1 | 27
  Male | 16 | 6 | 3 | 1 | 1 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 36 | 8 | 5 | 2 | 2 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 1 | 1 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 32 | 8 | 4 | 2 | 2 | 48
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1 and 2: Pharmacokinetics (PK) of Rilpivirine (TMC278) as Measured by Maximum Observed Plasma Concentration at Steady State (Cmax,ss)
Description: Cmax,ss was the maximum observed plasma concentration of rilpivirine at steady state (steady state starting from Day 14).
Time Frame: Pre-dose, 0, 2, 4, 5, 6, 9, 12 and 24 hours post dose at steady-state (any time during Day 14 to Day 18)
Population: Population: participants who took at least 1 dose of RPV, regardless of their compliance with protocol & adherence to dosing regimen. N (Overall number of participants analyzed) =participants evaluable for this outcome measure (OM). In this OM, summarized data for arms "Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg" and "Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg", is not reported as plan was to prepare & report participant wise data when "N" was <3 (which is reported in OM 2).
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 Children (>=25 kg): Rilpivirine 25 mg | Cohort 2 Children (<25 kg): Rilpivirine 25 mg
Number analyzed (Participants) | 23 | 6 | 4
nanograms per milliliter (ng/mL) | 109 (38.0) | 154 (52.2) | 238 (160)

2. Primary Outcome: Cohort 2: Pharmacokinetics (PK) of Rilpivirine (TMC278) as Measured by Maximum Plasma Concentration at Steady State (Cmax,ss)
Description: Cmax,ss was the maximum plasma concentration of rilpivirine at steady state (steady state starting from Day 14). In the below data table, the measure type "Number" corresponds to Cmax,ss concentration.
Time Frame: Pre-dose, 0, 2, 4, 5, 6, 9, 12 and 24 hours post dose at steady-state (any time during Day 14 to Day 18)
Population: Analysis population included all participants who had taken at least 1 dose of rilpivirine, regardless of their compliance with the protocol and adherence to the dosing regimen. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure. For this OM, participant wise data was only reported because individual data analysis was planned when the 'N' was less than 3.
Measure: Number; unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg | Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg
Number analyzed (Participants) | 2 | 2
nanograms per milliliter (ng/mL)
  Participant 1: number analyzed (Participants) | 1 | 0
  Participant 1 | 138 |
  Participant 2: number analyzed (Participants) | 1 | 0
  Participant 2 | 184 |
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 81.9
  Participant 4: number analyzed (Participants) | 0 | 1
  Participant 4 |  | 156

3. Primary Outcome: Cohorts 1 and 2: Pharmacokinetics of Rilpivirine as Measured by Area Under the Plasma Concentration Curve at Steady State (AUC24, ss)
Description: AUC24,ss was defined as the area under the plasma concentration versus time curve from time 0 to 24 hours post dosing of rilpivirine at steady state (steady state starting from Day 14).
Time Frame: Pre-dose, 0, 2, 4, 5, 6, 9, 12 and 24 hours post dose at steady-state (any time during Day 14 to Day 18)
Population: Population: participants who took at least 1 dose of RPV, regardless of their compliance with protocol & adherence to dosing regimen. N (Overall number of participants analyzed) = participants evaluable for this OM. In this OM, summarized data for arms "Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg" and "Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg", is not reported as plan was to prepare & report participant wise data when "N" was <3 (which is reported in OM 4).
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 Children (>=25 kg): Rilpivirine 25 mg | Cohort 2 Children (<25 kg): Rilpivirine 25 mg
Number analyzed (Participants) | 23 | 6 | 4
nanograms*hour per milliliter (ng*hr/mL) | 1872 (717) | 2610 (776) | 3339 (2233)

4. Primary Outcome: Cohort 2: Pharmacokinetics of Rilpivirine as Measured by Area Under the Plasma Concentration Curve at Steady State (AUC24, ss)
Description: AUC24,ss was defined as the area under the plasma concentration versus time curve from time 0 to 24 hours post dosing of rilpivirine at steady state (steady state starting from Day 14). In the below data table, the measure type "Number" corresponds to AUC24, ss concentration.
Time Frame: Pre-dose, 0, 2, 4, 5, 6, 9, 12 and 24 hours post dose at steady-state (any time during Day 14 to Day 18)
Population: as for outcome 2
Measure: Number; unit: ng*hr/mL
Arm/Group | Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg | Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg
Number analyzed (Participants) | 2 | 2
ng*hr/mL
  Participant 1: number analyzed (Participants) | 1 | 0
  Participant 1 | 1933 |
  Participant 2: number analyzed (Participants) | 1 | 0
  Participant 2 | 2877 |
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 1710
  Participant 4: number analyzed (Participants) | 0 | 1
  Participant 4 |  | 2958

5. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product and did not necessarily have a causal relationship with the treatment.
Time Frame: Cohort 1: From baseline (Day 1) up to Week 240; Cohort 2: From Baseline (Day 1) up to 240 weeks (for participants recruited up to protocol amendment 9); up to 48 weeks (for participants recruited after implementation of protocol amendment 10)
Population: Analysis population included all participants who had taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 Children (>=25 kg): Rilpivirine 25 mg | Cohort 2 Children (<25 kg): Rilpivirine 25 mg | Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg | Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg
Number analyzed (Participants) | 36 | 9 | 5 | 2 | 2
Participants | 35 | 8 | 5 | 2 | 2

6. Secondary Outcome: Cohorts 1 and 2: Percentage of Participants With Plasma Human Immunodeficiency Virus -1 (HIV-1) Ribonucleic Acid (RNA) Level Less Than (<) 50 Copies/mL by Time to Loss of Virologic Response (TLOVR) Method
Description: Percentage of participants with plasma HIV-1 RNA <50 copies per milliliter (Copies/mL) assessed by TLOVR method was reported. TLOVR requires sustained HIV-1 RNA < 50 copies/mL; confirmed HIV-1 RNA more than or equal to (>=) 50 copies/mL is considered as non-response (rebound); participant was considered non-responder after permanent discontinuation. Responder is defined as the participant with confirmed plasma viral load <50 copies/mL. As planned, combined data for cohort 2 was collected, analyzed and reported for this outcome measure.
Time Frame: At Week 48 (for Cohorts 1 and 2) and at Week 240 (for Cohort 1 only)
Population: Population: participants who took at least 1 dose of RPV, regardless of compliance with protocol & adherence to dosing regimen. In Cohort 2, "0" in "number analyzed" field of Week 240 = Week 240 was not applicable as it was beyond duration of Cohort 2 (Week 48); 0 in number analyzed field of Week 48 =planned TLOVR method was not used for data analysis per PA 10 and thus no data was reported in this OM. 'n' (number analyzed) =number of participants with available data at specified timepoints.
Measure: Number; unit: Percentage of participants
Groups:
- Cohort 2 (>=6 to <12 Years): Rilpivirine: Participants received rilpivirine tablet 25 mg or adjusted dose orally QD from baseline (Day 1) up to 240 weeks (for participants recruited up to protocol amendment 9); up to 48 weeks (for participants recruited after implementation of protocol amendment 10), in combination with an investigator-selected background regimen containing 2 N[t]RTIs: AZT, ABC, or TDF in combination with 3TC or FTC.
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 (>=6 to <12 Years): Rilpivirine
Number analyzed (Participants) | 36 | 0
Percentage of participants
  Week 48 | 72.2 |
  Week 240: number analyzed (Participants) | 32 | 0
  Week 240 | 43.8 |

7. Secondary Outcome: Cohorts 1 and 2: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/mL by Food and Drug Administration (FDA) Snapshot Approach
Description: Percentage of participants with a HIV-1 RNA <50 copies per mL were assessed using FDA snapshot approach which defines a participant's virologic response status using only the viral load at the predefined time point within a window of time, along with study drug discontinuation status. If HIV-1 RNA level is < 50 copies per mL, it is considered as virologic success as per the snapshot approach. As planned, combined data for cohort 2 was collected, analyzed and reported for this outcome measure.
Time Frame: At Week 48 (for Cohorts 1 and 2) and at Week 240 (for Cohort 1 only)
Population: Population:participants who took at least 1 dose of RPV, regardless of compliance with protocol & adherence to dosing regimen. "N"(Overall number of participants analyzed)=participants evaluable for this OM. "n"(number analyzed)=number of participants with available data at specified timepoints. In Cohort 2, '0' in 'number analyzed' at Week 240=Week 240 was beyond duration of Cohort 2 (Week 48). '0' in 'number analyzed' of Cohort 1 Week 48=snapshot method was not applicable for Cohort 1 Week 48.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 (>=6 to <12 Years): Rilpivirine
Number analyzed (Participants) | 32 | 18
Percentage of participants
  Week 48: number analyzed (Participants) | 0 | 18
  Week 48 |  | 72.2
  Week 240: number analyzed (Participants) | 32 | 0
  Week 240 | 53.1 |

8. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Post Baseline Genotype Data
Description: Number of participants with post baseline genotype (nucleoside analogue reverse transcriptase inhibitors [NRTI] and non-nucleoside reverse transcriptase inhibitors [NNRTI] resistance) data were reported. As planned, combined data for cohort 2 was collected, analyzed and reported for this outcome measure.
Time Frame: as for outcome 5
Population: Analysis population included all participants who had taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimen. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 (>=6 to <12 Years): Rilpivirine
Number analyzed (Participants) | 20 | 6
Participants
  NNRTI | 9 | 5
  NRTI | 7 | 4

9. Secondary Outcome: Cohorts 1 and 2: Percentage of Participants With Treatment Adherence >95% Based on Drug Accountability
Description: Percentage of participants with treatment adherence >95% based on drug accountability from baseline up to Week 240 for Cohort 1 and from baseline up to 240 weeks (for participants recruited up to protocol amendment 9); up to 48 weeks (for participants recruited after implementation of protocol amendment 10) for cohort 2 were reported. Treatment adherence was defined as having a treatment adherence of greater than (>) 95 percent (%) by pill count. Drug accountability included dispensation, receipt, and return, or if applicable, destruction of RPV documented by using the appropriate forms. As planned, combined data for cohort 2 was collected, analyzed and reported for this outcome measure.
Time Frame: as for outcome 5
Population: Analysis population included all participants who had taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimen. For Cohort 2, "0" in "number analyzed" field indicated that no participants were available for analysis at Week 240 for Cohort 2 arm because timepoint Week 240 was not applicable to Cohort 2 as it was beyond the duration of Cohort 2 (i.e., Week 48).
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 (>=6 to <12 Years): Rilpivirine
Number analyzed (Participants) | 36 | 18
Percentage of participants
  Up to 48 weeks | 80.6 | 77.8
  Up to 240 weeks: number analyzed (Participants) | 36 | 0
  Up to 240 weeks | 77.8 |

10. Secondary Outcome: Cohorts 1 and 2: Change From Baseline in Cluster of Differentiation (CD4+) Cells
Description: The immunologic change was determined by changes in Cluster of CD4+ cell count using non-completer =failure imputation, that is discontinuation was imputed with baseline value resulting in change=0, other missing data using last observation carried forward (LOCF). Change from baseline in CD4+ cell count at Week 48 for Cohort 1 and 2; and at Week 240 for Cohort 1 only were assessed. As planned, combined data for cohort 2 was collected, analyzed and reported for this outcome measure.
Time Frame: Baseline (Day 1) and Week 48 for Cohorts 1 and 2; Week 240 for Cohort 1 alone
Population: Analysis population included all participants who had taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimen. Here, 'n' (number analyzed) signifies the number of participants with available data at each specified timepoint. "0" participants in "number analyzed field" of cohort 2 indicated that Week 240 was not applicable to Cohort 2 as it was beyond the duration of Cohort 2 (i.e., Week 48).
Measure: Mean (Standard Error); unit: Cells per microliter
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 (>=6 to <12 Years): Rilpivirine
Number analyzed (Participants) | 36 | 18
Cells per microliter
  Week 48 | 201.2 (32.87) | 215.9 (62.42)
  Week 240: number analyzed (Participants) | 32 | 0
  Week 240 | 113.6 (26.72) |

ADVERSE EVENTS:
Time Frame: Cohort 1: From baseline (Day 1) up to Week 240; Cohort 2: From baseline (Day 1) up to 240 weeks (for participants recruited up to protocol amendment 9); up to 48 weeks (for participants recruited after implementation of protocol amendment 10)
Description: Analysis population included all participants who had taken at least 1 dose of rilpivirine, regardless of their compliance with the protocol and adherence to the dosing regimen.
  MedDRA 13.1 was used for Cohort 1 arm and MedDRA 25.0 was used for Cohort 2 arms.
Arm/Group | Cohort 1 Adolescents: Rilpivirine 25 mg | Cohort 2 Children (>=25 kg): Rilpivirine 25 mg | Cohort 2 Children (<25 kg): Rilpivirine 25 mg | Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg | Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/9 | 0/5 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 6/36 | 0/9 | 0/5 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 35/36 | 8/9 | 5/5 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Adolescents: Rilpivirine 25 mg (N=36) | Cohort 2 Children (>=25 kg): Rilpivirine 25 mg (N=9) | Cohort 2 Children (<25 kg): Rilpivirine 25 mg (N=5) | Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg (N=2) | Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg (N=2)
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Abscess Limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Suicide Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicidal Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Adolescents: Rilpivirine 25 mg (N=36) | Cohort 2 Children (>=25 kg): Rilpivirine 25 mg (N=9) | Cohort 2 Children (<25 kg): Rilpivirine 25 mg (N=5) | Cohort 2 Children (>=20 to <25 kg): Rilpivirine 15 mg (N=2) | Cohort 2 Children (<20 kg): Rilpivirine 12.5 mg (N=2)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0
Rheumatic Heart Disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 4 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 4 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Fungal Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 15 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 3 | 1 | 1 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 20 | 5 | 3 | 2 | 2
Urinary Tract Infection (Infections and infestations) | 4 | 0 | 0 | 0 | 0
Acth Stimulation Test Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 0 | 0 | 0 | 0
Blood Cortisol Decreased (Investigations) | 7 | 0 | 0 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Protein Total Increased (Investigations) | 2 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 4 | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 5 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 7 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 0 | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1
Tooth Extraction (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT00799864/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT00799864/SAP_001.pdf